CLINICAL TRIAL: NCT00925626
Title: Sub-Vastus Versus Mid-Vastus Arthrotomy for Total Knee Arthroplasty: a Randomized Clinical Trial With One Year Follow-up
Brief Title: Sub-Vastus Versus Mid-Vastus Arthrotomy for Total Knee Arthroplasty: a Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2009/256
Record Dates: First submitted 2009-06-19; First posted 2009-06-22 (Estimated); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Tricompartmental Gonarthrosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sub - Vastus arthrotomy (Experimental): Sub-vastus arthrotomy
  Interventions: Procedure: Sub-Vastus arthrotomy
- Mid-Vastus arthrotomy (Active Comparator): Mid-vastus arthrotomy
  Interventions: Procedure: Mid - Vastus arthrotomy

INTERVENTIONS:
Procedure: Sub-Vastus arthrotomy — Sub-vastus arthrotomy
  Arms: Sub - Vastus arthrotomy
Procedure: Mid - Vastus arthrotomy — Mid-vastus arthrotomy
  Arms: Mid-Vastus arthrotomy

SUMMARY:
Randomized, single-blind trial in which one group of patients will be operated with a "Mid-Vastus approach" of the knee joint and the other group will undergo knee surgery with a "Sub-Vastus approach".

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with osteoarthrosis of the knee
* patients must be in good general health condition

Exclusion Criteria:

* patients with morbid obesity (BMI >45)
* patients with history of knee surgery, infection or inflammatory disease of the knee joint or large cartilage lesion

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-06 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
VAS, KOOS and HSS scales | at day 1, day 2, day 3, day 4 and day 5 post-operatively
Rehabilitation time; time needed for 90° flexion of the knee joint | post-operatively

SECONDARY OUTCOMES:
VAS, HSS, KOOS questionnaires | at 6 weeks, 3 months and 12 months after surgery.
Amount and type of analgesic drugs used. | pre-operatively and post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Peter Verdonk, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: website of the University Hospital Ghent — http://www.uzgent.be